CLINICAL TRIAL: NCT01858428
Title: ILLUMENATE Pivotal: ProspectIve, Randomized, SingLe-Blind, U.S. MuLti-Center Study to EvalUate TreatMent of Obstructive SupErficial Femoral Artery or Popliteal LesioNs With A Novel PacliTaxel-CoatEd Percutaneous Angioplasty Balloon
Brief Title: Pivotal Trial of a Novel Paclitaxel-Coated Percutaneous Angioplasty Balloon
Acronym: ILLUMENATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TP-1397
Record Dates: First submitted 2013-05-08; First posted 2013-05-21 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bare PTA (Active Comparator): The control device is a commercially available PTA balloon catheter (EverCross™ 0.035 PTA Balloon Catheter, Covidien, Plymouth, MN 55441, USA).
  Interventions: Device: EverCross Percutaneous Transluminal Balloon Catheter
- Drug-Coated PTA (Experimental): The CVI Paclitaxel-coated PTA Catheter is a commercially available PTA balloon catheter (EverCross™ 0.035 PTA Balloon Catheter, Covidien, Plymouth, MN 55441, USA) coated with paclitaxel using a proprietary carrier.
  Interventions: Device: Cardiovascular Ingenuity (CVI) Paclitaxel-coated Percutaneous Transluminal Angioplasty Balloon Catheter

INTERVENTIONS:
Device: Cardiovascular Ingenuity (CVI) Paclitaxel-coated Percutaneous Transluminal Angioplasty Balloon Catheter — The CVI Paclitaxel-coated PTA Catheter is a commercially available PTA balloon catheter (EverCross™ 0.035 PTA Balloon Catheter, Covidien, Plymouth, MN 55441, USA) coated with paclitaxel using a proprietary carrier.
  Arms: Drug-Coated PTA
Device: EverCross Percutaneous Transluminal Balloon Catheter — The control device is a commercially available PTA balloon catheter (EverCross™ 0.035 PTA Balloon Catheter, Covidien, Plymouth, MN 55441, USA).
  Arms: Bare PTA

SUMMARY:
This study is designed to evaluate the safety and efficacy of a Paclitaxel-coated percutaneous transluminal angioplasty (PTA) Catheter in the treatment of patients with peripheral arterial disease.

DETAILED DESCRIPTION:
The ILLUMENATE Pivotal study is a prospective, randomized, multi-center, single-blind study which will include up to 360 subjects in approximately forty-five (45) sites across the United States to evaluate the CVI Paclitaxel-coated PTA Catheter compared to the bare percutaneous transluminal angioplasty balloon catheter (bare balloon catheter) for the treatment of de-novo or post-PTA occluded/stenotic or reoccluded/restenotic (except for in-stent) SFA and/or popliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with symptomatic leg ischemia, requiring treatment of the Superficial Femoral Artery (SFA) or popliteal artery.

Exclusion Criteria:

* Known intolerance to study medications, paclitaxel or contrast agents that in the opinion of the investigator cannot be adequately pre-treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-06-18 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Krishnan, MD, Principal Investigator — Mt. Sinai Medical Center; Sean Lyden, MD, Principal Investigator — The Cleveland Clinic
Locations (44):
- United States (42):
  - Yuma Regional Medical Center, Yuma, Arizona
  - Mission Cardiovascular Research Institute, Fremont, California
  - Good Samaritan Hospital - Los Angeles, Los Angeles, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Cardiovascular Research of North Florida, Gainesville, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Coastal Vascular and Interventional, Pensacola, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Advocate Health and Hospitals Corporation, Oakbrook Terrace, Illinois
  - St. Joseph Hospital, Fort Wayne, Indiana
  - Central Iowa Hospital Corporation, Des Moines, Iowa
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Mission Hospital, Asheville, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Wake Heart Research, Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - North Ohio Research LTD., Elyria, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Heritage Valley Health System, Beaver, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, INC., Wormleysburg, Pennsylvania
  - Providence Cardiology LLC, Columbia, South Carolina
  - Sanford Health Vascular Associates, Sioux Falls, South Dakota
  - University Surgical Associates, Chattanooga, Tennessee
  - Wellmont Holston Area Medical Center, Kingsport, Tennessee
  - Premier Surgical Associates, Knoxville, Tennessee
  - Texas Health & Research Education Institution, Dallas, Texas
  - El Paso Cardiology Associates, El Paso, Texas
  - University of Texas Health Science Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Sentara Vascular Specialist, Norfolk, Virginia
  - CAMC Clinical Trial Center, Charleston, West Virginia
  - Aurora Health Care, Milwaukee, Wisconsin
- Austria (2):
  - LKH Univ. - Klinikum Graz, Graz
  - Hanusch Krankenhaus Wien, Vienna

REFERENCES:
- [Derived] Krishnan P, Faries P, Niazi K, Sachar R, Jain A, Brodmann M, Werner M, Holden A, Tarricone A, Tarra T, Lyden S. Stellarex Drug-Coated Balloon for the Treatment of Peripheral Artery Disease: Five-Year Results from the ILLUMENATE Pivotal Randomized Controlled Trial. Am J Cardiol. 2024 Sep 15;227:83-90. doi: 10.1016/j.amjcard.2024.06.027. Epub 2024 Jul 15. PMID 39019203
- [Derived] Lyden SP, Brodmann M, Parikh SA, Krishnan P, Schroeder H, Werner M, Holden A, Ouriel K, Tarra T, Gray WA. Four-year patient-level pooled mortality analysis of the ILLUMENATE US Pivotal and EU randomized controlled trials. J Vasc Surg. 2022 Feb;75(2):600-607. doi: 10.1016/j.jvs.2021.07.244. Epub 2021 Sep 8. PMID 34506898
- [Derived] Gray WA, Jaff MR, Parikh SA, Ansel GM, Brodmann M, Krishnan P, Razavi MK, Vermassen F, Zeller T, White R, Ouriel K, Adelman MA, Lyden SP. Mortality Assessment of Paclitaxel-Coated Balloons: Patient-Level Meta-Analysis of the ILLUMENATE Clinical Program at 3 Years. Circulation. 2019 Oct;140(14):1145-1155. doi: 10.1161/CIRCULATIONAHA.119.040518. Epub 2019 Sep 30. PMID 31567024
- [Derived] Krishnan P, Faries P, Niazi K, Jain A, Sachar R, Bachinsky WB, Cardenas J, Werner M, Brodmann M, Mustapha JA, Mena-Hurtado C, Jaff MR, Holden AH, Lyden SP. Stellarex Drug-Coated Balloon for Treatment of Femoropopliteal Disease: Twelve-Month Outcomes From the Randomized ILLUMENATE Pivotal and Pharmacokinetic Studies. Circulation. 2017 Sep 19;136(12):1102-1113. doi: 10.1161/CIRCULATIONAHA.117.028893. Epub 2017 Jul 20. PMID 28729250

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization. Patients who provided written informed consent but were excluded from the study due to not meeting all of the inclusion criteria or meeting one or more of the exclusion criteria were screen failures. Subjects who had unsuccessful pre-dilatation were not randomized and were to be treated per the institution's standard of care.
Groups:
- Bare PTA: EverCross™ Balloon Catheter (PTA control device) (a product of Covidien during enrollment and now a product of Medtronic)
- Drug-Coated PTA: Cardiovascular Ingenuity (CVI) Paclitaxel-coated Percutaneous Transluminal Angioplasty Balloon Catheter: The CVI Paclitaxel-coated PTA Catheter is a commercially available PTA balloon catheter coated with paclitaxel using a proprietary carrier.
Period: Overall Study
Arm/Group | Bare PTA | Drug-Coated PTA
Started | 100 (EverCross™ Balloon Catheter now a product of Medtronic) | 200
Completed | 99 | 190
Not Completed | 1 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bare PTA | Drug-Coated PTA | Total
Number analyzed (Participants) | 100 | 200 | 300
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 69.8 (9.8) | 68.3 (10.3) | 68.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 88 | 124
  Male | 64 | 112 | 176
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Not all participants disclosed race or ethnicity.
  Participants
    American Indian or Alaska Native: number analyzed (Participants) | 96 | 190 | 286
    American Indian or Alaska Native | 0 | 2 | 2
    Asian: number analyzed (Participants) | 96 | 190 | 286
    Asian | 1 | 2 | 3
    Black or African American: number analyzed (Participants) | 96 | 190 | 286
    Black or African American | 19 | 35 | 54
    White: number analyzed (Participants) | 96 | 190 | 286
    White | 68 | 142 | 210
    Other: number analyzed (Participants) | 96 | 190 | 286
    Other | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  Austria | 10 | 17 | 27
  United States | 90 | 183 | 273
Ankle-Brachial Index [Mean (Standard Deviation); unit: ratio] — The ankle-brachial index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachium). The normal range for the ankle-brachial index is between 0.90 and 1.30. An index under 0.90 means that blood is having a hard time getting to the legs and feet: 0.41 to 0.90 indicates mild to moderate peripheral artery disease; 0.40 and lower indicates severe disease.
  ratio | 0.76 (0.20) | 0.75 (0.21) | 0.75 (0.21)
Rutherford Becker Clinical Category [Number; unit: participants] — Rutherford-Becker Classification is a classification system of Peripheral Arterial Disease, the higher the number the worse the disease.
  Category Clinical Description 0-Asymptomatic--no hemodynamically significant occlusive disease
  1. Mild claudication
  2. Moderate claudication
  3. Severe claudication 4*-Ischemic rest pain 5*-Minor tissue loss-nonhealing ulcer, focal gangrene with diffuse pedal ischemia 6*-Major tissue loss-extending above transmetatarsal level, functional foot no longer salvageable *Categories 4, 5, and 6 are also described as critical limb ischemia.
  participants
    Rutherford 2 | 35 | 63 | 98
    Rutherford 3 | 60 | 129 | 189
    Rutherford 4 | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Patency at 12 Month Post-procedure
Description: Patency is defined as the absence of target lesion restenosis as determined by duplex ultrasound (Peak Systolic Velocity Ratio (PSVR) ≤ 2.5) and freedom from clinically-driven target lesion revascularization.
Time Frame: 12 months
Population: Missing outcome status due to early study exit may differ from the total subjects exited by each visit interval as some subjects may have been eligible for failures carried forward or had a Clinically driven target lesion revasc (CD-TLR) prior to study exit.
Measure: Count of Participants; unit: Participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 92 | 177
Participants | 53 | 135

2. Primary Outcome: Freedom From Device and Procedure-related Death and Target Limb Major Amputation and Clinically-driven Target Lesion Revascularization
Description: Freedom from device and procedure-related death through 30 days post-procedure and freedom from target limb major amputation and clinically-driven target lesion revascularization through 12 months post-procedure.
Time Frame: 30 Days and 12 months
Population: Some Safety Status Missing at 12 Months Missing outcome status due to early study exit may differ from the total subjects exited by each visit interval as some subjects may have had a primary safety event within 12 months prior to study exit.
Measure: Count of Participants; unit: Participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 95 | 189
Participants | 79 | 174

3. Secondary Outcome: Major Adverse Event (MAE) Rate in the Hospital and at 1, 6, 12, 24, 36, 48 and 60 Months Post-procedure
Description: Major adverse event (MAE) rate in the hospital and at 1, 6, 12, 24, 36, 48 and 60 months post-procedure, defined as a composite rate of cardiovascular death, target limb major amputation and clinically-driven target lesion revascularization (TLR).
Time Frame: 1, 6, 12, 24, 36, 48 and 60 months
Measure: Number; unit: Events
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 96 | 191
Events | 17 | 18

4. Secondary Outcome: Rate of Vascular Access and Bleeding Complications
Description: Rate of vascular access and bleeding complications in the hospital and at 1, 6, 12 and 24 months.
Time Frame: in-hospital and 1, 6, 12 and 24 months
Measure: Number; unit: participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 95 | 190
participants | 3 | 8

5. Secondary Outcome: Rate of Clinically-driven Target Lesion Revascularization
Time Frame: 6, 12, 24, 36, 48 and 60 months
Measure: Number; unit: participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 95 | 189
participants | 15 | 16

6. Secondary Outcome: Rate of Target Lesion Revascularization
Time Frame: 6, 12, 24, 36, 48 and 60 months
Measure: Number; unit: participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 95 | 189
participants | 17 | 18

7. Secondary Outcome: Rate of Target Limb Major Amputation
Time Frame: 1, 6, 12, 24, 36, 48 and 60 months
Measure: Number; unit: participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 95 | 189
participants | 0 | 0

8. Secondary Outcome: Mortality Rate
Time Frame: 6, 12, 24, 36, 48 and 60 months
Measure: Number; unit: participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 96 | 192
participants | 2 | 5

9. Secondary Outcome: Rate of Occurrence of Arterial Thrombosis of the Treated Segment
Time Frame: 1, 6, 12, 24, 36, 48 and 60 months
Measure: Number; unit: participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 95 | 189
participants | 0 | 2

10. Secondary Outcome: Patency Rate and Freedom From Clinically-driven TLR
Description: Patency rate defined as the absence of target lesion restenosis as determined by duplex ultrasound (PSVR ≤ 2.5) and freedom from clinically-driven TLR at 6, 24 and 36 months
Time Frame: 6, 24 and 36 months
Measure: Number; unit: participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 84 | 152
participants | 58 | 133

11. Secondary Outcome: Lesion Success of Achieving a Final In-lesion Residual Diameter Stenosis of ≤50%
Description: Lesion success, defined as achievement of a final in-lesion residual diameter stenosis of ≤50% (as determined by the angiographic core lab), using any device after wire passage through the lesion.
Time Frame: procedure, Day 0
Measure: Number; unit: participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 100 | 199
participants | 98 | 196

12. Secondary Outcome: Technical Success of Achieving a Final In-lesion Residual Diameter Stenosis of ≤50%
Description: Technical success, defined as achievement of a final in-lesion residual diameter stenosis of ≤50% (as determined by the angiographic core lab), using the CVI Paclitaxel-coated PTA Catheter or bare balloon catheter without a device malfunction after wire passage through the lesion.
Time Frame: procedure, Day 0
Measure: Number; unit: Lesion
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 100 | 199
Lesion | 98 | 196

13. Secondary Outcome: Per Subject Clinical Success Achieving no Major Adverse Events During the Procedure
Description: Clinical success (per subject) defined as technical success without the occurrence of major adverse events during the procedure.
Time Frame: procedure, Day 0
Measure: Number; unit: participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 100 | 199
participants | 98 | 196

14. Secondary Outcome: Per Subject Procedural Success Achieving no Major Adverse Events During the Procedure
Description: Procedural success (per subject) defined as lesion success without the occurrence of major adverse events during the procedure.
Time Frame: procedure, Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 100 | 199
Participants | 98 | 196

15. Secondary Outcome: Change in Ankle-brachial Index (ABI) From Pre-procedure
Description: Subjects who had reinterventions were included in ABI analyses so some improvements may be reflective of revascularizations during the follow-up period.
Time Frame: 6, 12, 24 and 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bare PTA | Drug-Coated PTA
Number analyzed (Participants) | 91 | 167
Participants | 69 | 132

ADVERSE EVENTS:
Time Frame: 12 months
Description: Events are stratified by MedDRA system organ class (SOC) and preferred term (PT). Subjects may experience multiple event types, thus the sum of the subjects by PT need not equal the total number of subjects in the summary for each SOC. In cases where the event verbatim term was updated by the Clinical Events Committee (CEC), the MedDRA coding was based on the event verbatim term provided by the CEC. Otherwise, the MedDRA coding was based on the site-reported event verbatim term.
Arm/Group | Bare PTA | Drug-Coated PTA
All-Cause Mortality (participants affected / at risk) | 2/100 | 5/200
Serious Adverse Events (participants affected / at risk) | 63/100 | 120/200
Other Adverse Events (participants affected / at risk) | 85/100 | 162/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bare PTA (N=100) | Drug-Coated PTA (N=200)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 3 (4)
Angina Pectoris (Cardiac disorders) | 2 (3) | 5 (7)
Angina Unstable (Cardiac disorders) | 1 (1) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 4 (4)
Atrioventricular Block (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 2 (6)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 3 (4)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 3 (3)
Sick Sinus Syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Blindness Unilateral (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Retinal Artery Occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's Oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Angiodysplasia Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Intestinal Ischaemia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter Site Haematoma (General disorders) | 0 (0) | 1 (1)
Catheter Site Haemorrhage (General disorders) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 1 (1)
Chest Pain (General disorders) | 4 (4) | 8 (12)
Death (General disorders) | 2 (2) | 0 (0)
Device Occlusion (General disorders) | 0 (0) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 2 (2)
Sudden Cardiac Death (General disorders) | 0 (0) | 1 (1)
Vessel Puncture Site Thrombosis (General disorders) | 0 (0) | 1 (1)
Bile Duct Stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis Perforated (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (3)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bursitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (3) | 2 (2)
Diabetic Foot Infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
H1N1 Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 2 (3)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 4 (5)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral Arterial Reocclusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 7 (8) | 8 (8)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasm Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Artery Stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 6 (6)
Renal Failure Chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Obesity Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral Revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Toe Amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Wound Drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Aortic Stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Femoral Artery Dissection (Vascular disorders) | 6 (6) | 17 (17)
Femoral Artery Occlusion (Vascular disorders) | 0 (0) | 1 (2)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 4 (4)
Intermittent Claudication (Vascular disorders) | 6 (6) | 16 (17)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 3 (3)
Peripheral Artery Dissection (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Stenosis (Vascular disorders) | 18 (21) | 22 (23)
Peripheral Embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1) | 3 (3)
Venous Insufficiency (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bare PTA (N=100) | Drug-Coated PTA (N=200)
Chest Pain (General disorders) | 6 (6) | 14 (20)
Oedema Peripheral (General disorders) | 5 (5) | 7 (7)
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 11 (13) | 12 (12)
Arthralagia (Musculoskeletal and connective tissue disorders) | 10 (10) | 14 (14)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 12 (12)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (11)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 13 (13) | 24 (30)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 10 (10)
Femoral Artery Dissection (Vascular disorders) | 6 (6) | 17 (19)
Intermittent Claudication (Vascular disorders) | 17 (19) | 33 (49)
Peripheral Artery Stenosis (Vascular disorders) | 26 (34) | 31 (39)

LIMITATIONS AND CAVEATS:
Per FDA confirmation letter, dated April 10, 2018, Re: G120270/R012, this study concluded March 19, 2018. Subjects rolled into the post-approval study (NCT03421561). Long-term follow-up data can be found there for remaining study objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days